CLINICAL TRIAL: NCT06848660
Title: Rigid Collar or No Collar for Non-surgical Treatment of Stable Cervical Spine Fractures: a Protocol for a Randomized Register Trial
Brief Title: Study on Orthosis in Cervical Spine Fracture Treatment
Acronym: SOFT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Anna Mac Dowall, Associate Professor, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOFT
Record Dates: First submitted 2025-02-20; First posted 2025-02-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Cervical Spine Fractures; Cervical Spine Injury; Rigid Collar
Keywords: cervical spine fracture treatment; cervical rigid collar; rigid collar treatment; subaxial fractures; odontoid fractures

STUDY DESIGN:
Intervention Model Description: The SOFT is a nationwide, multicenter, open label, cluster randomized crossover Register-RCT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-surgical treatment with a rigid collar (Experimental): Non-surgical treatment with a rigid collar The patient will be recommended to wear a rigid collar at all times, and to be careful, for 12 weeks. The choice of supplier and brand of the cervical collar is decided by the treatment guidelines in each hospital. No planned return visits are planned for the intervention-group. The clinical routine for patients receiving non-surgical treatment is a follow-up with a fracture control including a CT scan at 10-14 days after the trauma. Physiotherapy and other rehabilitation measures will be considered and prescribed on an individual basis.
  Interventions: Device: A rigid cervical collar
- Non-surgical treatment without a rigid collar (No Intervention): The patient will be recommended to be careful, for 12 weeks but will otherwise have no specified restrictions. The patients will follow the same clinical routine regarding a follow-up with a fracture control including a CT scan at 10-14 days after the trauma. Physiotherapy and other rehabilitation measures will be considered and prescribed on an individual basis.

INTERVENTIONS:
Device: A rigid cervical collar — The rigid cervical collar is used for spinal motion restriction for 12 weeks for the non-surgical treatment of a stable cervical spine fracture.
  Arms: Non-surgical treatment with a rigid collar

SUMMARY:
Background and Purpose:

Neck fractures affect over 1,100 people in Sweden each year, with the majority being frail older adults. Most neck fractures are stable and therefore treated without surgery, typically using a rigid collar. However, the collar only limits neck movement by 40-50% and can cause pressure sores, as well as difficulties with swallowing and breathing. Because of these issues, the latest Swedish national guidelines for pre-hospital and hospital spinal motion restriction have replaced the rigid collar with other methods. This raises the question of whether the rigid collar still has a role in the modern treatment of stable neck fractures.

The aim of this study is to determine whether treatment with or without a rigid collar leads to equally good healing outcomes.

Method:

All adults diagnosed with a stable neck fracture deemed suitable for non-surgical treatment will be included in the study at the time of registration in the Swedish Fracture Register (SFR). Participating hospitals will be randomly assigned (1:1) to either use no collar at all or a rigid collar for 12 weeks. After an initial period of 1.5 years, the hospitals will switch to the opposite treatment group. A total of 616 participants are expected to be included within 3 years.

At the one-year follow-up, investigators will evaluate how many participants in each treatment group that required a switch to surgical stabilization due to treatment failure. Secondary outcomes will include quality of life, neck pain, and the need for assistive devices in relation to disability and complications in both groups.

Summary:

Non-surgical treatment rarely fails, and the need to switch from non-surgical treatment to surgery is very uncommon. The rigid collar is often prescribed out of habit, without much consideration for its potential negative effects. If this study shows that the rigid collar is unnecessary for treating stable neck fractures, frail older adults-who often struggle with collar-related discomfort, malnutrition, and pressure sores-could avoid unnecessary suffering.

DETAILED DESCRIPTION:
The annual incidence rate of spinal fracture is 64 per 100,000 with a peak in young men and elderly women (1). Ten percent of all traumatic spinal fractures are located in the upper cervical spine and 20% in the subaxial cervical spine (2). Stable cervical spine fractures are treated non-surgically, with a rigid collar that is worn 24 hours a day for 12 weeks to limit neck movements and promote bone healing. However, rigid collars only restrict 40-50% of cervical spine motions (3, 4). The drawbacks with collar treatment are that the collar may be very uncomfortable, may cause pressure ulcer, or affect swallowing or breathing (5). Wearing a collar is associated with difficulties to perform activities of daily living due to the limited neck movement. Treatment without a collar would avoid the annoyance and potential harm, whilst the stable fracture may still heal.

Investigators aim to compare the benefit versus the harm and discomfort of rigid collar treatment with treatment without a rigid collar, in a registry based randomized controlled trial.

Treatment decisions may be made using a fracture classification such as the Subaxial injury classification and severity scale (SLICS) (6) or others. C1 and C2 fractures have separate classifications. In C1 fractures a lateral dislocation of > 7 mm is classified as unstable and requires surgical fixation. In the elderly, C2 fractures are common, secondary to low energy trauma and are mostly regarded as stable (7).

Cervical spine fractures are common enough to be a significant public health problem but too uncommon to perform a prospective study comparing the results of current treatments in a single institution. Quality registers are excellent alternatives to close these knowledge gaps. The Swedish fracture register (SFR) is a national register founded in 2011. Spinal fractures have been included since 2015, and the intra- and interrater reliability is acceptable (8). The diagnosing physician classifies the fracture with the help of drawings.

Treatment, non-surgical, or surgical treatment is registered as well as treatment failure, non-surgical treatment converted to surgical stabilization and secondary surgery after failure of the primary surgery. Patient reported outcome measures (PROMs) are sent to the participants shortly after the fracture occurrence (concerning status before the injury), and at one-year of follow-up. The PROMs include the European quality of life 5 dimensions 5 level (EQ-5D-5L) (9) and the Short Musculoskeletal Function Assessment (SMFA) (10). In SFR the treatment failure on cervical spine fractures treated non-surgically is 4% and the most common cause of failure is patients with facet joint dislocation or anterior distraction with posterior compression (manuscript in preparation). However, facet joint dislocation and anterior distraction do not often fall within the recommendations of non-surgical treatment. Investigators consider it to be safe conducting this trial. Investigators expect essentially none of the participants assigned to non-surgical treatment with or without a rigid collar to face the risk of undergoing surgical treatment.

In clinicaltrials.gov there are 3 registered trials on rigid collars; 1) The DENS trial comparing early removal versus 12 weeks treatment with a rigid collar in older frail adults with odontoid fractures (NCT04895644) (11), 2) A pilot efficacy trial comparing parathyroid hormone analog (PTH) together with a rigid collar versus historical treatment with rigid collar alone (NCT04760782), 3) A study about the length of rigid collar treatment, 6 versus 12 weeks (NCT02788760). Two randomized controlled trials (RCT) compare surgical versus non-surgical treatment of odontoid fractures in the elderly (NCT03788200, NCT02789774).

Considering the rigid collars limited effectiveness on spinal motion restriction and the potential harm they may afflict there is reason to explore the additional value of rigid collars in non-surgical treatment of stable cervical spine fractures, compared with no use of rigid collars.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged > 18 years with a stable cervical spine fracture*.
* A history of recent trauma (within 3 weeks).
* Recruited within 3 weeks of injury.
* Determined by the consultant spinal surgeon as suitable for non-surgical treatment.

Exclusion Criteria:

* New neurological deficit attributable to the fracture.
* Additional cervical spine fracture not suitable for non-surgical treatment.
* Underlying condition with risk of spinal instability (e.g., ankylosing spondylitis, DISH, rheumatoid arthritis).
* Fracture suspected to be older than 3 weeks at the time of assessment.
* Not expected to survive to hospital discharge or not expected to survive surgical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants that had surgery within 1 year after the fracture incident | From enrollment to the 1 year of follow-up
  Treatment failure, defined as non- surgical treatment converted to surgical treatment, measured at 1 year of follow-up. All participants that receive cervical spine surgery within 1 year after the cervical spine fracture incident, are accounted for and compared between the groups.

SECONDARY OUTCOMES:
European quality of life 5 dimensions 5 lite (EQ-5D 5L) | From enrollment to 1 year of follow-up.
  Change from baseline to one year of follow-up, in the EQ-5D 5L index with a higher number representing better life quality, ranging from -0.59 to 1.00 (10).
European quality of life health scale (EQ-5D health) | From enrollment to 1 year of follow-up.
  Change from baseline to one year of follow-up, in EQ-5D health, ranging from 0-100 with higher scores indicating better health.
Short musculoskeletal function assessment (SMFA) | From enrollment to 1 year of follow-up.
  Change from baseline to one year of follow-up, in the SMFA (11), a 46-item questionnaire describing the patient´s musculoskeletal function, containing both a dysfunction index and a bother index. The indexes range from 0-100.
Adverse events | From enrollment to 1 year of follow-up.
  Adverse events might be pressure ulcer, difficulty in swallowing or breathing or other uncomfortable experiences. Prolonged neck pain and fracture pseudarthrosis is an adverse event as long as no surgical treatment has been performed to resolve the neck pain or fracture pseudarthrosis.
Mortality | From enrollment to 1 year of follow-up.
  The participant has deceased.

OTHER OUTCOMES:
Neck disability index (NDI) | From enrollment to 1 year of follow-up.
  A subgroup analysis will be performed to investigate the disability in participants following a cervical spine fracture. One of the most common disease specific indices for neck pain and disability is the NDI (16). NDI ranges from 0-100 % with higher scores indicating severe disability. The MCID is 15%-17% (16, 17). NDI is not available in the Swedish fracture register, while the EQ-5D and SMFA is. A subgroup of 100 participants in Uppsala will be asked to fill in both NDI and the SMFA to investigate correlations between the two PROMs. Our previous experience is that the Oswestry disability index (ODI), the corresponding disability index constructed for back pain, have a high correlation to SMFA (18). It is likely that NDI has a similar correlation to SMFA as ODI.
Compliance to rigid collar treatment | From enrollment to 12 weeks of follow-up.
  A single-center sub-group of 50 patients will be asked to participate in a study concerning compliance to rigid collar treatment. After verbal and written information and a signed consent has been obtained a small sensor will be placed inside the cervical collar. The sensor measures the warmth from the neck when the collar is worn and will register if the collar is taken off.
Osteopororsis screening | From enrollment to 12 weeks of follow-up.
  A single-center sub-group of 50 participants with a stable cervical spine fracture assigned to non-surgical treatment, will be asked to participate in a study concerning osteoporosis screening. After verbal and written information and a signed consent has been obtained, a Dual energy X-ray Absorptiometry (DXA) will be performed. If the participant already has been screened with a DXA previously a new DXA will examine the change in bone mineral density (BMD) over time.

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized data and the R code used for statistical analysis may be shared upon request after the final publication of the results of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Pseudonymized data and the R code used for statistical analysis may be shared upon request after the final publication of the results of the study.
Access Criteria: The data will only be shared for the sake of study reproducibility. Upon a request stated to the principal investigator a data sharing agreement must be agreed upon and signed. The GDPR officer at Uppsala University Hospital will help setting up the data sharing agreement according to laws and regulations. Data sharing outside the European Union cannot be guaranteed at this date.
  After signed agreement, pseudonymized data and the R code might be securely transferred by a software with a secure 2 stage verification.

REFERENCES:
- [Background] Blixt S, Mukka S, Forsth P, Westin O, Gerdhem P; SunBurst study group. Study protocol: The SunBurst trial-a register-based, randomized controlled trial on thoracolumbar burst fractures. Acta Orthop. 2022 Jan 24;93:256-263. doi: 10.2340/17453674.2022.1614. PMID 35175357
- [Background] Woodfield J, Edlmann E, Black PL, Boyd J, Copley PC, Cranswick G, Eborall H, Keerie C, Khan S, Lawton J, Lowe DJ, Norrie J, Niven A, Reed MJ, Shenkin SD, Statham P, Stoddart A, Tomlinson J, Brennan PM. Duration of External Neck Stabilisation (DENS) following odontoid fracture in older or frail adults: protocol for a randomised controlled trial of collar versus no collar. BMJ Open. 2022 Jul 15;12(7):e057753. doi: 10.1136/bmjopen-2021-057753. PMID 35840308
- [Background] Swiontkowski MF, Engelberg R, Martin DP, Agel J. Short musculoskeletal function assessment questionnaire: validity, reliability, and responsiveness. J Bone Joint Surg Am. 1999 Sep;81(9):1245-60. doi: 10.2106/00004623-199909000-00006. PMID 10505521
- [Background] Burstrom K, Teni FS, Gerdtham UG, Leidl R, Helgesson G, Rolfson O, Henriksson M. Experience-Based Swedish TTO and VAS Value Sets for EQ-5D-5L Health States. Pharmacoeconomics. 2020 Aug;38(8):839-856. doi: 10.1007/s40273-020-00905-7. PMID 32307663
- [Background] Morgonskold D, Warkander V, Savvides P, Wihlborg A, Bouzereau M, Moller H, Gerdhem P. Inter- and intra-rater reliability of vertebral fracture classifications in the Swedish fracture register. World J Orthop. 2019 Jan 18;10(1):14-22. doi: 10.5312/wjo.v10.i1.14. eCollection 2019 Jan 18. PMID 30705837
- [Background] Koivikko MP, Kiuru MJ, Koskinen SK, Myllynen P, Santavirta S, Kivisaari L. Factors associated with nonunion in conservatively-treated type-II fractures of the odontoid process. J Bone Joint Surg Br. 2004 Nov;86(8):1146-51. doi: 10.1302/0301-620x.86b8.14839. PMID 15568528
- [Background] Vaccaro AR, Hulbert RJ, Patel AA, Fisher C, Dvorak M, Lehman RA Jr, Anderson P, Harrop J, Oner FC, Arnold P, Fehlings M, Hedlund R, Madrazo I, Rechtine G, Aarabi B, Shainline M; Spine Trauma Study Group. The subaxial cervical spine injury classification system: a novel approach to recognize the importance of morphology, neurology, and integrity of the disco-ligamentous complex. Spine (Phila Pa 1976). 2007 Oct 1;32(21):2365-74. doi: 10.1097/BRS.0b013e3181557b92. PMID 17906580
- [Background] Peck GE, Shipway DJH, Tsang K, Fertleman M. Cervical spine immobilisation in the elderly: a literature review. Br J Neurosurg. 2018 Jun;32(3):286-290. doi: 10.1080/02688697.2018.1445828. Epub 2018 Feb 28. PMID 29488398
- [Background] Whitcroft KL, Massouh L, Amirfeyz R, Bannister GC. A comparison of neck movement in the soft cervical collar and rigid cervical brace in healthy subjects. J Manipulative Physiol Ther. 2011 Feb;34(2):119-22. doi: 10.1016/j.jmpt.2010.12.007. PMID 21334544
- [Background] The Effectiveness of Four Contemporary Cervical Orthoses in Restricting Cervical Motion Lunsford, Thomas R. MSE, CO; Davidson, Michael; Lunsford, Brenda R. MAPT, MS Author Information JPO Journal of Prosthetics and Orthotics 6(4):p 93-99, Fall 1994.
- [Background] Tee JW, Chan CH, Fitzgerald MC, Liew SM, Rosenfeld JV. Epidemiological trends of spine trauma: an Australian level 1 trauma centre study. Global Spine J. 2013 Jun;3(2):75-84. doi: 10.1055/s-0033-1337124. Epub 2013 Mar 19. PMID 24436855
- [Background] Hu R, Mustard CA, Burns C. Epidemiology of incident spinal fracture in a complete population. Spine (Phila Pa 1976). 1996 Feb 15;21(4):492-9. doi: 10.1097/00007632-199602150-00016. PMID 8658254